CLINICAL TRIAL: NCT06396091
Title: A Phase 1 Open-label Study to Assess the Safety and Tolerability of Zolbetuximab (IMAB362) in Combination With Chemotherapy (mFOLFIRINOX) in Participants With CLDN18.2 Positive Metastatic Pancreatic Adenocarcinoma
Brief Title: A Study of Zolbetuximab With Chemotherapy in Adults With Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8951-CL-5203
Expanded Access: NCT06048081 (Available)
Record Dates: First submitted 2024-04-30; First posted 2024-05-02 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: CLDN18.2 positive metastatic pancreatic adenocarcinoma; mFOLFIRINOX; Claudin 18.2
MeSH Terms: interventions — zolbetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- zolbetuximab and mFOLFIRINOX (Experimental): Participants will receive 1 of 2 dose levels of zolbetuximab in combination with mFOLFIRINOX.
  Interventions: Drug: zolbetuximab; Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: zolbetuximab — Zolbetuximab will be administered intravenously on day 1 then every two weeks.
  Other Names: IMAB362
Drug: mFOLFIRINOX — Modified oxaliplatin, leucovorin, irinotecan and fluorouracil (mFOLFIRINOX) will be administered intravenously within 2 days after administration of zolbetuximab.

SUMMARY:
Pancreatic cancer is difficult to diagnose early. By the time people have been diagnosed, the cancer has usually spread to other parts of the body (metastatic). The standard treatment is chemotherapy, but other treatments are needed to improve outcomes in people with pancreatic cancer.

In this study, zolbetuximab will be given together with chemotherapy to people with pancreatic cancer. Zolbetuximab attaches to a protein called CLDN18.2 found at high levels on the surface of the cancer tumor. This switches on the immune system to attack the tumor.

Adults 18 years or older with metastatic pancreatic cancer who have not previously had chemotherapy can take part in the study.

There are 2 main aims of this study:

* To check the safety of zolbetuximab, when given with chemotherapy in people with metastatic pancreatic cancer
* To check if people could cope with (tolerate) any medical problems during the study This is an open-label study. This means people in the study and the study doctors will know that people will receive zolbetuximab with chemotherapy. Different small groups will receive lower to higher doses of zolbetuximab with chemotherapy.

Zolbetuximab and chemotherapy will be given through a vein. This is called an infusion. People will receive zolbetuximab on the first day they receive chemotherapy. This will happen every 14 days in a 28-day cycle.

People will receive zolbetuximab and chemotherapy in the study clinic and at home. Also, doctors will check for any medical problems. People will also have a health check including blood tests. On some visits they will also have scans to check for any changes in their cancer.

People will visit the study clinic about 7 days after they stop treatment. They will be asked about any medical problems and will have a health check including blood tests.

After this, people will have several more visits to the study clinic for health checks. The number of visits and checks done at each visit will depend on the health of each person and whether they complete their treatment or not.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically or cytologically confirmed adenocarcinoma of pancreas.
* Participant must have metastatic pancreatic adenocarcinoma that has not been previously treated with chemotherapy:

  * Prior treatment with 5-fluorouracil or gemcitabine administered as a radiation sensitizer during and up to 4 weeks after radiation therapy is allowed (if there is lingering toxicity, then the sponsor should be consulted).
  * If a participant received neoadjuvant/adjuvant therapy, tumor recurrence or disease progression must have occurred at least 6 months after completing the last dose of the neoadjuvant/adjuvant therapy.
  * Participant whose disease progressed on prior treatment with mFOLFIRINOX are not eligible.
* Participant has a measurable lesion(s) on at least 1 metastatic site based on RECIST v1.1 within 28 days prior to enrollment. For participants with only 1 measurable lesion and prior radiotherapy, the lesion must be outside the field of prior radiotherapy or must have documented progression following radiation therapy.
* Participant's tumor is CLDN18.2 positive, defined as ≥ 75% of tumor cells demonstrating moderate to strong membranous CLDN18 staining as determined by central immunohistochemistry testing.
* Female subject is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who has a negative urine or serum pregnancy test at screening or within 48 hours prior to day 1; and agrees to follow the contraceptive guidance from the time of informed consent through through 9 months after the final administration of oxaliplatin and 6 months after the final administration of all other study interventional drugs.
* Female participant must not be breastfeeding or lactating starting at screening and throughout the treatment period and for 6 months after the final study intervention administration.
* Female participant must not donate ova starting at first administration of study intervention and throughout the treatment period and for 6 months after the final study intervention administration.
* A male participant must agree to use contraception with female partner(s) of childbearing potential (including breastfeeding partner) throughout the treatment period and for 6 months after final study intervention administration.
* A male participant must agree to remain abstinent or use a condom with pregnant partner(s) for the duration of the pregnancy throughout the treatment period and for 6 months after final study intervention administration.
* A male participant must not donate sperm during the treatment period and for 6 months after final study intervention administration.
* Participant agrees not to participate in another interventional study while receiving study intervention in the present study/participating in the present study.
* Participant has ECOG performance status 0 or 1.
* Participant has predicted life expectancy ≥ 12 weeks.
* Participant must meet all of the following criteria based on the laboratory tests collected within 14 days prior to enrollment. In case of multiple laboratory data within this period, the most recent data should be used.
* Participant must meet all of criteria based on laboratory tests during screening period.

Exclusion Criteria:

* Participant has prior severe allergic reaction; suspected, known immediate or delayed hypersensitivity; or intolerance or contraindication to known ingredients of zolbetuximab or other monoclonal antibody, including humanized or chimeric antibodies.
* Participant has prior severe allergic reaction; suspected, known immediate or delayed hypersensitivity; or intolerance or contraindication to any component of mFOLFIRINOX.
* Participant has known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Participant has a known history of a positive test for human immunodeficiency virus infection or known active hepatitis B (positive HBs Ag) or hepatitis C infection.

  * For participants who are negative for hepatitis B surface antigen, but hepatitis B core antibody positive, a hepatitis B virus deoxyribonucleic acid test will be performed and if positive, the participant will be excluded.
  * Participants with positive hepatitis C serology but negative hepatitis C virus ribonucleic acid test results are eligible.
  * Participants treated for hepatitis C with undetectable viral load results are eligible.
* Participant has a history of interstitial pneumonia or pulmonary fibrosis.
* Participant has pleural effusion or ascites ≥ Grade 3 per Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
* Participant has an active autoimmune disease that has required systemic treatment in the past 3 months prior to enrollment.
* Participant has active infection requiring systemic therapy that has not completely resolved within 7 days prior to enrollment.
* Participant has significant cardiovascular disease, including:

  * Congestive heart failure (defined as New York Heart Association Class III or IV), myocardial infarction, unstable angina, coronary angioplasty, coronary stenting,coronary artery bypass graft, cerebrovascular accident or hypertensive crisis within 6 months prior to enrollment;
  * History of clinically significant ventricular arrhythmias (i.e., sustained ventricular tachycardia, ventricular fibrillation or torsades de pointes);
  * QT interval corrected for heart rate (QTc) > 450 msec for male participants; QTc interval > 470 msec for female participants;
  * Cardiac arrhythmias requiring anti-arrhythmic medications (Participants with rate-controlled atrial fibrillation for > 1 month prior to enrollment are eligible).
* Participant has a history of central nervous system metastases and/or carcinomatous meningitis from pancreatic adenocarcinoma.
* Participant has known peripheral sensory neuropathy ≥ Grade 2 per CTCAE v5.0 unless the absence of deep tendon reflexes is the sole neurological abnormality.
* Participant has had diarrhea within 24 hours prior to enrollment.
* Participant has had a major surgical procedure ≤ 28 days prior to enrollment.
* Participant without complete recovery from a major surgical procedure ≤ 14 days prior to enrollment.
* Participant has a psychiatric illness or social situations that would preclude study compliance.
* Participant has another malignancy for which treatment is required.
* Participant has any concurrent disease, infection or co-morbid condition that interferes with the ability of the participant to participate in the study, which places the participant at undue risk or complicates the interpretation of data.
* Participant has received radiotherapy for metastatic pancreatic adenocarcinoma unless the radiotherapy was completed > 14 days prior to enrollment and has recovered from any related toxicity.
* Participant has received systemic immunosuppressive therapy, including systemic corticosteroids within 14 days prior to enrollment.
* Participant using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg per day of hydrocortisone or up to 10 mg per day of prednisone), receiving a single dose of systemic corticosteroids or receiving systemic corticosteroids as premedication for radiologic imaging contrast use is allowed.
* Participant has a present or previous history of participation in a study of the study intervention.
* Participant has a previous history of investigational study intervention administration.
* Participant uses strong inhibitors or inducers of CYP3A or UGT1A1 when using irinotecan.
* Participant has received any investigational therapy within 28 days prior to screening.
* Participant has any condition which makes the participant unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLT) | Up to 28 days
  A DLT will be defined as any event meeting the DLT criteria occurring during the DLT assessment period that is related to zolbetuximab.
Safety assessed by Adverse Events (AEs) | Up to 16 months
  An AE is any untoward medical occurrence in a patient or clinical study participant temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator, if applicable, and events related to the (study) procedures.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to 16 months
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or adverse events (AEs) | Up to 16 months
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiograms (ECG) abnormalities and or adverse events | Up to 16 months
  Number of participants with potentially clinically significant ECG values.
Number of participants at each grade of Eastern Cooperative Oncology Group (ECOG) performance status scores | Up to 15 months
  The ECOG scale will be used to assess performance status. Grades range from 0 (fully active) to 5 (dead). Negative change scores indicate an improvement. Positive scores indicate a decline in performance.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of zolbetuximab in serum: End of infusion concentrations | Up to 1 month
  End of infusion concentrations will be derived from the PK serum samples collected.
PK of zolbetuximab in serum: Concentration Immediately Prior to Dosing at multiple dosing (Ctrough) | Up to 12 months
  Ctrough will be derived from the PK serum samples collected.
Number of participants with positive antidrug antibodies (ADA) to zolbetuximab | Up to 15 months
Change from baseline in Cancer Antigen 19-9 (CA 19-9) | Baseline up to 13 months
  Serum CA19-9 will be assessed.
Best Overall Response (BOR) Rate | Up to 15 months
  The BOR is determined once all tumor response data for the participant is available. Participants will be classified by BOR on study as outlined in Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Overall Response Rate (ORR) | Up to 15 months
  ORR is defined as the proportion of participants with best overall response as confirmed complete response (CR) or partial response based on RECIST v1.1 as assessed by investigator.
Disease Control Rate (DCR) | Up to 15 months
  DCR is defined as the proportion of participants with a complete or partial response as assessed by investigator based on RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.